CLINICAL TRIAL: NCT02915588
Title: Early Active Rehabilitation After Arthroscopic Rotator Cuff Repair: A Prospective Randomized Pilot Study
Brief Title: Early Active Rehabilitation After Arthroscopic Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Kepler University of Linz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PMR-Shoulder-001
Record Dates: First submitted 2016-09-15; First posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Full Thickness Rotator Cuff Tear

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Primary Active (Active Comparator): Early postoperative isometric activation of the rotator cuff
  Interventions: Other: early isometric loading after rotator cuff surgery
- Primary Passive (Active Comparator): Standard postoperative passive movement rehabilitation protocol
  Interventions: Other: passive motion after rotator cuff surgery

INTERVENTIONS:
Other: early isometric loading after rotator cuff surgery
  Arms: Primary Active
Other: passive motion after rotator cuff surgery
  Arms: Primary Passive

SUMMARY:
The purpose of the study is to compare two different rehabilitation protocols after arthroscopic rotator cuff surgery.

ELIGIBILITY:
Inclusion Criteria:

* surgery of the rotator cuff after full thickness tear
* informed consent
* understanding german language

Exclusion Criteria:

* previous surgery of the shoulder
* neurological or systemic diseases with impairment of shoulder function

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change of Constant Murley Score | up to 24 weeks
  Timepoints: Before surgery; 6, 12, 24 weeks after surgery

SECONDARY OUTCOMES:
Change of DASH Score | up to 24 weeks
  Timepoints Before surgery; 6, 12, 24 weeks after surgery
Change of Active range of Motion (Flexion, Extension, Abduction, Internal Rotation, External Rotation) | up to 24 weeks
  Timepoints: Before surgery; 6, 12, 24 weeks after surgery; Range of movement is measured by handheld goniometer
Change of Pain (max; average; rest) | up to 24 weeks
  Timepoints: Before surgery; 6, 12, 24 weeks after surgery; Pain is measured by Visual Analogue Scale (0-100mm)
Change of Strength (abduction; external Rotation) | up to 24 weeks
  Timepoints: Before surgery; 6, 12, 24 weeks after surgery; Measurement of Strength is evaluated using a BTE Simulator II Dynamometer (Peak torque in N).

CONTACTS AND LOCATIONS:
Overall Officials: Christian Mittermaier, Dr, Principal Investigator — Institute of physical medicine and rehabilitation
Locations (1):
- Kepler University Hospital, Linz, Austria

IPD SHARING:
Plan to Share IPD: No